CLINICAL TRIAL: NCT07252102
Title: Effect of High Flow Nasal Cannula Oxygenation on Incidence of Hypoxia During Sedated Gastrointestinal Endoscopy in Critical Patients: A Multicentre Randomised Controlled Trial
Brief Title: Effect of HFNC on Incidence of Hypoxia During Sedated Gastrointestinal Endoscopy in Critical Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Diansan Su, Chief, Department of Anesthesiology, the First Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZJU2025C036
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Liver Cirrhosis; Polyps of Colon; Gastrointestinal Dysfunction
Keywords: critical patients; HFNC; High flow nasal cannulas oxyge; hypoxia
MeSH Terms: conditions — Liver Cirrhosis; Colonic Polyps; Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flow nasal catheter oxygen (Experimental)
  Interventions: Device: High-flow nasal catheter oxygen
- Regular nasal catheter oxygen (Active Comparator)
  Interventions: Device: regular nasal catheter oxygen

INTERVENTIONS:
Device: High-flow nasal catheter oxygen — Before induction of anesthesia, connect the Airvo2 (HFNC high flow device) special nasal cannula to inhale oxygen, and preoxygenate with an oxygen flow rate of 6L /min. After induction of anesthesia, adjust the oxygen flow rate to 60L /min, oxygen concentration 100%, oxygen temperature 37℃ until the end of gastrointestinal endoscopy.
  Arms: High-flow nasal catheter oxygen
Device: regular nasal catheter oxygen — Before anesthesia induction, a disposable nasal catheter oxygen inhalation device (covered by HFNC nasal catheter and blinded to the patient) was connected to an oxygen source for pre-oxygen inhalation, 6L/min. After induction of anesthesia, oxygen was continued for 6L/min until the end of gastroenteroscopy.
  Arms: Regular nasal catheter oxygen

SUMMARY:
High flow nasal cannula oxygenation (HFNC) offers high flow and concentration oxygen delivery, providing excellent non-respiratory oxygenation. As a relatively new oxygen delivery method, it has gained widespread use. We have demonstrated that high flow nasal cannula oxygenation reduce the incidence of hypoxia during sedated gastrointestinal endoscopy in patients with American Anesthesiologist Rating (ASA rating) grades 1 to 2 and obesity. We hypothesized that HFNC could mitigate the risk of hypoxia in critical patients during sedated gastrointestinal endoscopy. To confirm this, we selected critical patients with ASA grades 3 to 4 who were scheduled for gastrointestinal endoscopy. We observed and compared the incidence of hypoxia (75%≤SpO2 < 90% and < 60S), severe hypoxia (SpO2<75% for any duration or 75%≤SpO2 < 90%, ≥60s), subclinical respiratory depression (90%≤SpO2 < 95%), respiratory-related adverse events, sedation-related adverse events, and complications associated with high flow nasal cannula oxygenation using HFNC or regular nasal cannula during the sedated gastrointestinal endoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. 18≤ age ≤80, gender is not limited;
2. Patients undergoing elective gastroenteroscopy or treatment;
3. ASA grade Ⅲ~Ⅳ;
4. 18 kg/m2≤BMI≤28kg/m2;
5. The operation time of gastroenteroscopy is expected to be no more than 60min;
6. Clearly understand, voluntarily participate in the study, and have informed consent from myself or my family members.

Exclusion Criteria:

1. Patients with nasal congestion, nasal bleeding, recent nasal trauma, recent nasal surgery, increased intracranial pressure and skull fracture, etc., who can not perform high-flow nasal catheter oxygen;
2. acute respiratory infections and asthma attacks;
3. Patients diagnosed with COPD;
4. Clear difficult airway;
5. Acute upper gastrointestinal bleeding with shock;
6. Gastrointestinal obstruction with gastric content retention;
7. Allergic to sedatives such as propofol;
8. Persons with no capacity for civil conduct such as cognitive dysfunction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  75%≤ SpO2 < 90% and < 60S

SECONDARY OUTCOMES:
Incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  SpO2<75% for any duration, or 75%≤SpO2 < 90%, ≥60s
Incidence of subclinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  90%≤ SpO2<95%

OTHER OUTCOMES:
The incidence of other adverse events | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided